CLINICAL TRIAL: NCT01826188
Title: Combined THC and CBD Drops for Treatment of Crohn's Disease, a Phase II Double Blind Placebo Controlled Trial
Brief Title: Combined THC and CBD Drops for Treatment of Crohn's Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0196-12-MMC
Record Dates: First submitted 2013-03-28; First posted 2013-04-08 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; IBD Cannabis; THC; CBD
MeSH Terms: conditions — Crohn Disease | interventions — Dronabinol; Cystathionine beta-Synthase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- THC 5 mg/ml and CBD 50 mg/ml. (Active Comparator): olive oil containing THC 5 mg/ml and CBD 50 mg/ml. which will be taken twice daily.
  Interventions: Drug: THC 5mg/ml and CBS 50mg/ml
- Placebo (Placebo Comparator): olive oil but without any active ingredients.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC 5mg/ml and CBS 50mg/ml — olive oil containing THC and CBD
  Arms: THC 5 mg/ml and CBD 50 mg/ml.
Drug: Placebo — olive oil without cannabis
  Arms: Placebo

SUMMARY:
There are many reports about efficacy of Cannabis in Crohn's disease but no controlled trials. The aim of the proposed trial is to investigate the efficacy of oil containing the cannabinoids THC and CBD given by mouth for induction of remission in Crohn's disease.

DETAILED DESCRIPTION:
The investigators have recently published a retrospective observational study about the beneficial effect of cannabis in Crohn's disease. The investigators have also concluded a double blind placebo controlled study of Inhaled cannabis in the treatment of Crohn's disease. Both studies have shown significant symptomatic improvement of disease. However, objective parameters of inflammation were not measured. The question arises as to whether the observed improvement is merely symptomatic or due to a real change in inflammation. In addition, administration per os is a healthier option than smoking but the efficacy of oral cannabis was not investigated.

The aim of the proposed study in to evaluate the efficacy of drops of cannabis oil in crohn's disease patients compared to placebo. Treatment success will be defined as a decrease of at least 100 points in CDAI after 8 weeks of treatment.

Secondary aims:

1. Remission of disease i.e CDAI of less the 150 points.
2. Improvement of at least one point in Endoscopic disease activity index
3. Improvement of CRP and calprotectine
4. Improvement of blood cytokine levels
5. Improvement of at least 30 points in quality of life as measured by the SF 36. In addition the investigators will monitor side effects by questionnaires addressed to the patients and to a significant relative of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of Crohn's disease of at least 3 months duration, which was proved by either endoscopy or appropriate imaging study.
2. Patients who have failed treatment with either 5 ASA or corticosteroids or immunomodulators or biologic agents, or steroid dependant patients, or patients who were treated by the above mentioned drugs and could not tolerate them due to side effects.
3. Age 20 or older.
4. Able to sign informed concent
5. Active Crohn's disease with a CDAI 200 or more.

   -

Exclusion Criteria:

1. Patients with a diagnosis of a mental disorder
2. Patients who by the judgment of their physician are likely to develop drug addiction.
3. Pregnant women or women who are intending to become pregnant
4. Patients with a known cannabis allergy
5. Patients who are not capable of giving an informed consent
6. Patients with an impending operation due to Crohn's disease.

   -

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-03; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Treatment sucsess will be defind as a decrease of at least 100 points in CDAI after 8 weeks of treatment. | 8 weeks
  The aim of the proposed study in to evaluate the efficacy of drops of cannabis oil in crohn's diseas patients compared to placebo. Treatment sucsess will be defind as a decrease of at least 100 points in CDAI after 8 weeks of treatment.

SECONDARY OUTCOMES:
Remission of disease | 8 weeks
  1. Remission of disease i.e CDAI of less the 150 points.
endoscopic improvment | 8 week
  2. Improvment of at least one point in Endoscopic disease activity index
Improvment of CRP and calprotectine | 8 week
  CRP and calprotectine will be measured before and after 8 weeks of study treatment
Improvment of blood cytokine levls | 8 weeks
  blood cytokine levls including IL-10, TNF, and IL 23 will be measured before and at the end of the study
Improvment of at least 30 points in quality of life as measured by the SF 36. | 8 weeks
  patients will answer a short form of Health related quality of life quasionnair before and at the end of the study.

OTHER OUTCOMES:
Safety and side effects | 8 weeks
  we will monitor side effects by questionnairs adressed to the patients and to a significant relative of the patients.both patient and a significant realitive (parent, spouse) living in the same residence with the patient will recive a quationnair monitiring cannabis use, with aminimus score of 0 (not dependant, no side effects) to a maximum score of 15 (very dependant, sever side effects)

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Hospital, Kfar Saba, Israel

REFERENCES:
- [Background] Naftali T, Lev LB, Yablecovitch D, Half E, Konikoff FM. Treatment of Crohn's disease with cannabis: an observational study. Isr Med Assoc J. 2011 Aug;13(8):455-8. PMID 21910367